CLINICAL TRIAL: NCT01028495
Title: A Dose Tolerability and Efficacy Study of RX-0201 Plus Gemcitabine in Metastatic Pancreatic Cancer
Brief Title: A Safety and Efficacy Study of RX-0201 Plus Gemcitabine in Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rexahn Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RX-0201-P2-A-07
Record Dates: First submitted 2009-12-07; First posted 2009-12-09 (Estimated); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Metastatic Pancreatic Cancer
Keywords: AKT-1
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — RX-0201; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- gemcitabine and RX-0201 (Experimental): Gemcitabine at 1000 mg/day once a week for a 4 week cycle; 3 weeks of treatment at 30 minutes infusion once a week and one week off.
  RX-0201 3 week cycle at 250mg/m2/day of continuous infusion for 14 days with 7 days off.
  Interventions: Drug: RX-0201 plus Gemcitabine

INTERVENTIONS:
Drug: RX-0201 plus Gemcitabine — RX-0201 3 week cycle at 250mg/m2/day of continuous infusion for 14 days with 7 days off. Gemcitabine at 1000 mg/day once a week for a 4 week cycle; 3 weeks of treatment at 30 minutes infusion once a week and one week off.

SUMMARY:
To assess the safety and efficacy of a combined therapy regimen of RX-0201 plus Gemcitabine, in subjects with metastatic pancreatic cancer.

DETAILED DESCRIPTION:
Subjects enrolled to assess safety will receive a combination of Gemcitabine plus RX-0201. Gemcitabine will be administered prior to RX-0201 intravenously in a 30-min iv infusion dose at 1000 mg/m2 once weekly for up to 2 cycles; each 4-week cycle consist of 3-week treatment phase followed by 1 week resting phase. RX-0201 will be administered at 250 mg/m2/day in a 24-hour continuous intravenous infusion for up to 2 cycles; each 3-week cycle consists of 2-week treatment phase followed by a 1 week resting phase. (See schedule of assessments)Subjects enrolled to evaluate efficacy will receive a combination of Gemcitabine and RX-0201 as outline above for up to 4 cycles.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent prior to the initiation of study procedures.
* Are > 18 years of age
* Have metastatic pancreatic cancer.
* Have at least 1 measurable lesion by RECIST criteria.
* Have a Karnofsky Performance Status of > 70.
* Have at least a 6-month life expectancy as assessed by the investigator.
* Pre-menopausal women must be surgically sterile or agree to use an accepted method of birth control while participating in the study and for 30 days following the last exposure of study drug. Acceptable forms of birth control are: hormonal contraceptives (oral, injectable, transdermal or implant), double-barrier contraceptives (condom or diaphragm with spermicide), and intrauterine device (IUD).
* Male subjects need to either be surgically sterile or agree to use a barrier method of birth control described above during the study and for 30 days following the last exposure to study drug. The subject's agreed upon method of birth control will be discussed and documented in the subjects source document during the screening phase of the study.

Exclusion Criteria:

* Are unwilling or unable to provide informed consent.
* Are unwilling or unable to comply with the requirements of the protocol.
* Have been treated with another investigational agent for pancreatic cancer.
* Have any of the following screening laboratory values:

  * Hemoglobin < 8.0 grams/deciliter (g/dL)
  * Absolute neutrophil count (ANC) < 1500/microliter (μL)
  * Platelet count < 100,000/μL
  * Serum creatinine > 1.5 x the institutional upper limit of normal (IULN) creatinine.
  * Serum bilirubin > 1.5 X IULN
  * Aspartate transaminase (AST) (serum glutamic oxaloacetic transaminase, SGOT) > 2 x IULN (> 5 x IULN in presence of known liver metastasis)
  * Alanine transaminase (ALT) (serum glutamate pyruvate transaminase, SGPT) > 2 x IULN (> 5 x IULN in presence of known liver metastasis)
  * Have a prothrombin time >1.25 x IULN on screening laboratory assessments.
  * HCV or HBsAg positive subjects
* Have received therapeutic dose of either warfarin or heparin within 21 days before Day 1 (the first day of dosing; prophylactic use of warfarin or heparin) to maintain patency of indwelling IV catheters/lines is allowed
* Have a history of brain cancer (primary or metastatic).
* Have a history of an active hematologic malignancy within the past 2 years.
* Have an underlying diagnosis or disease state associated with an increased risk of bleeding (i.e., coagulopathies, HIV).
* Have a serious infection requiring intravenous antibiotic therapy during screening.
* Females who are pregnant, lactating, or have a positive serum pregnancy test during the screening period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2009-05; Primary Completion 2012-07 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Survival | 7 Months

SECONDARY OUTCOMES:
Tumor Response | 8 weeks assessment and 16 weeks to confirm
Toxicity and Safety Parameters | Continuously
Karnofsky Performance Scale, Clinical Laboratory Assessment, and Molecular Markers | Every 14 Days and Study Completion

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Tempero, M.D, Study Chair
Locations (10):
- United States (4):
  - Baptist Cancer Institute, Jacksonville, Florida
  - Orchard Healthcare Research Inc., Skokie, Illinois
  - Texas Oncology, Austin, Texas
  - Texas Oncology, P.A., McAllen, Texas
- India (6):
  - Jawaharlal Nehru Cancer Hospital and Research Centre, Bhopal, Kerala
  - Meenakshi Mission Hospital and Research Center, Madurai-625020
  - Central India Cancer Research Institute, Maharashtra
  - Shatabdi Superspeciality Hospital, Maharashtra
  - Rajiv Gandhi Cancer Institute and Research Center, Rohini New- Delhi
  - King George Hospital, Visakhapatanam, A.P

REFERENCES:
- [Background] Yoon H, Kim DJ, Ahn EH, Gellert GC, Shay JW, Ahn CH, Lee YB. Antitumor activity of a novel antisense oligonucleotide against Akt1. J Cell Biochem. 2009 Nov 1;108(4):832-8. doi: 10.1002/jcb.22311. PMID 19693774
- [Result] Journal of Clinical Oncology, 2007 ASCO Annual Meeting Proceedings Part I. Vol 25, No. 18S (June 20 Supplement), 2007: 3564